CLINICAL TRIAL: NCT06838585
Title: Intra-Abdominal Sepsis in Critically Ill Surgical Patients: the Relationship Between Cumulative Fluid Balance and Serum Sodium and Chloride Levels and In-Hospital Mortality
Brief Title: Intra-Abdominal Sepsis and Relationship Between Cumulative Fluid Balance and Serum Sodium and Chloride Levels and In-Hospital Mortality
Status: Completed | Type: Observational
Sponsor: Clinical Center of Vojvodina (Other)
Responsible Party: Principal Investigator, Radmila Nedeljko Popovic, Assistant Professor, Clinical Center of Vojvodina
Other Study IDs: 00-108
Record Dates: First submitted 2025-02-10; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Intraabdominal Infections; Fluid Balance; Disorder; Sodium Disorder; Chloride Disorder
Keywords: sepsis; intra-abdominal sepsis; in-hospital mortality; fluid therapy; sodium disorder; chloride disorder; critically ill patients
MeSH Terms: conditions — Intraabdominal Infections; Sepsis | interventions — Home Infusion Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: infusion therapy — Monitoring patients with fluid overload and fluid accumulation

SUMMARY:
Intra-abdominal sepsis and septic shock in critically ill surgical patients have a high mortality rate. Fluid therapy is one of the initial resuscitation measures, but it can contribute to poor treatment outcomes through fluid overload and accumulation of sodium and chloride. This study aimed to examine an association among cumulative fluid balance and serum sodium and chloride levels in the intensive care unit (ICU) and in-hospital mortality in critically ill surgical patients with intra-abdominal sepsis after emergency surgical treatment. The study was designed as a retrospective, cohort study.

DETAILED DESCRIPTION:
Data were collected and analyzed from 100 critically ill surgical patients with intra-abdominal sepsis, consecutively admitted to the ICU of a university medical center. Patients were immediately subjected to surgical treatment for intra-abdominal sepsis upon hospital admission. Postoperative care continued in the ICU for at least seven days. Patients who were hospitalized in the ICU for less than seven days, immunocompromised, and patients with intra-abdominal sepsis as a result of previous abdominal surgery were not included in the study. Data related to daily fluid intake and loss were taken from medical records where these data are recorded daily. Intake included both enteral and parenteral, while fluid losses from the body included urine, losses through drains, and nasogastric tube. The cumulative fluid balance was calculated for the periods from days 1 to 3 of treatment, and from days 1 to 7 of treatment. Data on serum sodium and chloride levels were recorded at the same time points as for cumulative fluid balance. The impact of variables on treatment outcomes was determined using binary logistic regression. The predictive quality of the variables on the outcome was assessed using ROC curves.

ELIGIBILITY:
Inclusion Criteria:

* critically ill surgical patients with intra-abdominal sepsis/septic shock consecutively admitted to a university medical center
* Patients who were immediately subjected to surgical treatment for intra-abdominal sepsis/sepstic shock upon hospital admission and postoperative care continued in the ICU for at least seven days

Exclusion Criteria:

* Patients who were hospitalized in the ICU for less than seven days
* immunocompromised
* patients with intra-abdominal sepsis as a result of previous abdominal surgery were not included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 critically ill surgical patients with intra-abdominal sepsis, consecutively admitted to the ICU of a university medical center. Patients were immediately subjected to surgical treatment for intra-abdominal sepsis upon hospital admission. Postoperative care continued in the ICU for at least seven days.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Association among cumulative fluid balance and serum sodium and chloride levels in the intensive care unit (ICU) and in-hospital mortality in critically ill surgical patients with intra-abdominal sepsis after emergency surgical treatment. | 2 years
  This study aimed to examine an association among cumulative fluid balance and serum sodium and chloride levels in the intensive care unit (ICU) and in-hospital mortality in critically ill surgical patients with intra-abdominal sepsis after emergency surgical treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Radmila N Popovic, MD, PhD, Principal Investigator — University Clinical Center of Vojvodina
Locations (1):
- Clinical Center of Vojvodina, Novi Sad, Serbia, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Popovic R, Andelic N, Jovanovic G, Maricic Prijic S, Uvelin A, Tomic N, Plecas Ethuric A, Todorovic N, Milijasevic B, Markovic D. Intra-abdominal sepsis in critically ill surgical patients: the relationship between cumulative fluid balance and serum sodium and chloride levels and in-hospital mortality. Front Med (Lausanne). 2025 Jul 16;12:1608388. doi: 10.3389/fmed.2025.1608388. eCollection 2025. PMID 40740943